CLINICAL TRIAL: NCT00174343
Title: Phase II Study Evaluating The Role Of Exemestane On Clinical And Pathologic Response Rates, And Its Aromatase Activity As Treatment In Neoadjuvant Setting For Operable Breast Cancer Patients.
Brief Title: Exemestane As Treatment In Neoadjuvant Setting For Operable Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 971-ONC-0028-095
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane

INTERVENTIONS:
Drug: exemestane (Aromasin®)

SUMMARY:
To evaluate clinical and pathologic response rates following primary hormonal therapy by exemestane (Aromasin®)

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal patients with unilateral breast cancer T2 to T4, N0-1, M0, non inflammatory, operable, hormonal receptors positive

Exclusion Criteria:

* Patients with bilateral breast cancer T4d, inflammatory, non operable, hormonal receptors negative

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46
Dates: Start 2001-11; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical and pathologic response rates following primary hormonal therapy by exemestane (Aromasin®)

SECONDARY OUTCOMES:
To evaluate breast conservative surgery rate; To evaluate intratumoral anti-aromatase activity.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- France (5):
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Saint-Cloud

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=971-ONC-0028-095&StudyName=Exemestane+As+Treatment+In+Neoadjuvant+Setting+For+Operable+Breast+Cancer+Patients